CLINICAL TRIAL: NCT01705145
Title: A Phase 3, 2-Part, Open-Label Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Ivacaftor in Subjects With Cystic Fibrosis Who Are 2 Through 5 Years of Age and Have a CFTR Gating Mutation
Brief Title: Study of Ivacaftor in Cystic Fibrosis Subjects 2 Through 5 Years of Age With a CFTR Gating Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-770-108; KIWI
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ivacaftor (Experimental): Part A: Ivacaftor 50 milligram (mg) (for participants weighing less than [<] 14 kilograms [kg]) or 75 mg (for participants weighing greater than or equal to [>=] 14 kg) every 12 hours (q12h) from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study..
  Part B: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h for 24 weeks during Part B of the study.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor
  Other Names: Kalydeco; VX-770

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD), of ivacaftor in children with cystic fibrosis (CF) who are 2 through 5 years of age and have a CF Transmembrane Conductance Regulator (CFTR) gating mutation in at least 1 allele.

Part A is designed to evaluate the safety and PK of multiple-dose administration of ivacaftor in participants 2 through 5 years of age and to confirm the doses for Part B. Part B is designed to evaluate the safety, PK, PD, and efficacy of ivacaftor in participants 2 through 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF
* Must have a CFTR gating mutation in at least 1 allele
* Aged 2 through 5 years at screening and Day 1
* Weight >= 8 kg at screening and Day 1
* Hematology, serum chemistry, coagulation, and vital signs results at screening with no clinically significant abnormalities that would interfere with the study assessments, as judged by the investigator

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* An acute upper or lower respiratory infection, or pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks before Day 1
* Abnormal liver function, at screening
* History of solid organ or hematological transplantation
* Use of any moderate or strong inducers or inhibitors of cytochrome P450 (CYP) 3A within 2 weeks before Day 1
* Participation in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 terminal half-lives before screening

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rosenfeld, MD, Principal Investigator — Seattle Children's Hospital; Jane Davies, MD, Principal Investigator — Imperial College London
Locations (20):
- United States (16):
  - Birmingham, Alabama
  - Aurora, Colorado
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Vancouver, Canada
- United Kingdom (3):
  - Edinburgh
  - Liverpool
  - London

REFERENCES:
- [Derived] Davies JC, Cunningham S, Harris WT, Lapey A, Regelmann WE, Sawicki GS, Southern KW, Robertson S, Green Y, Cooke J, Rosenfeld M; KIWI Study Group. Safety, pharmacokinetics, and pharmacodynamics of ivacaftor in patients aged 2-5 years with cystic fibrosis and a CFTR gating mutation (KIWI): an open-label, single-arm study. Lancet Respir Med. 2016 Feb;4(2):107-15. doi: 10.1016/S2213-2600(15)00545-7. Epub 2016 Jan 21. PMID 26803277

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivacaftor: Part A: Ivacaftor 50 milligram (mg) (for participants weighing less than [<] 14 kilograms [kg]) or 75 mg (for participants weighing greater than or equal to [>=] 14 kg) every 12 hours (q12h) from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study.
  Part B: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h for 24 weeks during Part B of the study. Part B included participants from Part A and newly enrolled participants.
Period: Part A
Arm/Group | Ivacaftor
Started | 9
Completed | 9
Not Completed | 0
Period: Part B
Arm/Group | Ivacaftor
Started | 34 (Eight participants from Part A continued in Part B of the study.)
Completed | 33
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of study drug.
Groups:
- Ivacaftor: Part A: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study.
  Part B: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h for 24 weeks during Part B of the study. Part B included participants from Part A and newly enrolled participants.
Arm/Group | Ivacaftor
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies participants who were evaluable for specified part of the study.
  years
    Part A (n = 9) | 3.1 (1.17)
    Part B (n = 34) | 3.2 (0.96)
Sex/Gender, Customized [Number; unit: participants] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies participants who were evaluable for specified part of the study.
  participants
    Part A (n = 9): Female | 3
    Part A (n = 9): Male | 6
    Part B (n = 34): Female | 6
    Part B (n = 34): Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Related AEs
Description: AE: any adverse change from participant's baseline (pre-treatment) condition, including any adverse experience, abnormal recording/clinical laboratory assessment which occurs during course of study, whether it is considered related to study drug or not. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event.
  Related AEs includes all AEs for which the causality was either related to study drug or possibly related to study drug. Data was reported as per the dose received and for overall participants.
Time Frame: Part A: Up to 93 Days
Population: Part A Safety set included all participants who received at least 1 dose of study drug in part A.
Measure: Number; unit: participants
Groups:
- Part A: Ivacaftor 50 mg: Ivacaftor 50 mg (for participants weighing <14 kg) q12h from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study.
- Part A: Ivacaftor 75 mg: Ivacaftor 75 mg (for participants weighing >=14 kg) q12h from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study.
- Part A: Overall Ivacaftor: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h from Day 1 through Day 3 and 1 morning dose on Day 4 during Part A of the study.
Arm/Group | Part A: Ivacaftor 50 mg | Part A: Ivacaftor 75 mg | Part A: Overall Ivacaftor
Number analyzed (Participants) | 4 | 5 | 9
participants
  AEs | 3 | 5 | 8
  SAEs | 0 | 0 | 0
  Related AEs | 1 | 3 | 4

2. Primary Outcome: Part B: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Related AEs
Description: AE: any adverse change from participant's baseline (pre-treatment) condition, including any adverse experience, abnormal recording/clinical laboratory assessment which occurs during course of study, whether it is considered related to study drug or not. AE includes both serious and non-serious AE. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event.
  Related AEs includes all AEs for which the causality was either related to study drug or possibly related to study drug. Data was reported as per the dose received.
Time Frame: Part B: Up to 28 Weeks
Population: Part B Safety set included all participants who received at least 1 dose of study drug in part B.
Measure: Number; unit: participants
Groups:
- Part B: Ivacaftor 50 mg: Ivacaftor 50 mg (for participants weighing <14 kg) q12h for 24 weeks during Part B of the study. Part B included participants from Part A and newly enrolled participants.
- Part B: Ivacaftor 75 mg: Ivacaftor 75 mg (for participants weighing >=14 kg) q12h for 24 weeks during Part B of the study. Part B included participants from Part A and newly enrolled participants.
- Part B: Overall Ivacaftor: Ivacaftor 50 mg (for participants weighing <14 kg) or 75 mg (for participants weighing >=14 kg) q12h for 24 weeks during Part B of the study. Part B included participants from Part A and newly enrolled participants.
Arm/Group | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Number analyzed (Participants) | 10 | 24 | 34
participants
  AEs | 10 | 23 | 33
  SAEs | 3 | 3 | 6
  Related AEs | 3 | 8 | 11

3. Secondary Outcome: Part B: Plasma Concentration of Ivacaftor and Its Metabolites
Description: Plasma concentration was reported for ivacaftor and its metabolites (M1 and M6) up to 24 hours post-dose on Day 168 (Hour 0 [predose] on Day 1, 14, 56, 112, and 168; 2, 3, 6 hours post-dose on Day 14; 1 hour post-dose on Day 56; 4, 6 hours post-dose on Day 112; 24 hours post-dose on Day 168). Data was planned to be reported for overall participants in the period.
Time Frame: Part B: up to 24 hours post-dose on Day 168
Population: Part B Safety set included all participants who received at least 1 dose of study drug in part B.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: Overall Ivacaftor
Number analyzed (Participants) | 34
ng/mL
  Ivacaftor: Hour 0 on Day 1 | 0.00 (0.00)
  Ivacaftor: Hour 0 on Day 14 | 614 (590)
  Ivacaftor: 2 Hours Post-Dose on Day 14 | 932 (541)
  Ivacaftor: 3 Hours Post-Dose on Day 14 | 1080 (587)
  Ivacaftor: 6 Hours Post-Dose on Day 14 | 1140 (627)
  Ivacaftor: Hour 0 on Day 56 | 448 (455)
  Ivacaftor: 1 Hour Post-Dose on Day 56 | 514 (421)
  Ivacaftor: Hour 0 on Day 112 | 596 (747)
  Ivacaftor: 4 Hours Post-Dose on Day 112 | 1080 (835)
  Ivacaftor: 6 Hours Post-Dose on Day 112 | 1010 (885)
  Ivacaftor: Hour 0 on Day 168 | 500 (545)
  Ivacaftor: 24 Hours Post-Dose on Day 168 | 207 (372)
  M1: Hour 0 on Day 1 | 0.00 (0.00)
  M1: Hour 0 on Day 14 | 1580 (1030)
  M1: 2 Hours Post-Dose on Day 14 | 1870 (924)
  M1: 3 Hours Post-Dose on Day 14 | 2280 (1140)
  M1: 6 Hours Post-Dose on Day 14 | 2670 (1080)
  M1: Hour 0 on Day 56 | 1340 (880)
  M1: 1 Hour Post-Dose on Day 56 | 1170 (698)
  M1: Hour 0 on Day 112 | 1680 (1360)
  M1: 4 Hours Post-Dose on Day 112 | 2450 (1510)
  M1: 6 Hours Post-Dose on Day 112 | 2500 (1520)
  M1: Hour 0 on Day 168 | 1460 (1200)
  M1: 24 Hours Post-Dose on Day 168 | 602 (647)
  M6: Hour 0 on Day 1 | 0.00 (0.00)
  M6: Hour 0 on Day 14 | 1520 (1130)
  M6: 2 Hours Post-Dose on Day 14 | 1430 (989)
  M6: 3 Hours Post-Dose on Day 14 | 1630 (1130)
  M6: 6 Hours Post-Dose on Day 14 | 2090 (1350)
  M6: Hour 0 on Day 56 | 1510 (1080)
  M6: 1 Hour Post-Dose on Day 56 | 1310 (974)
  M6: Hour 0 on Day 112 | 1660 (1130)
  M6: 4 Hours Post-Dose on Day 112 | 1810 (1230)
  M6: 6 Hours Post-Dose on Day 112 | 2130 (1380)
  M6: Hour 0 on Day 168 | 1520 (1130)
  M6: 24 Hours Post-Dose on Day 168 | 632 (465)

4. Secondary Outcome: Part B: Absolute Change From Baseline in Sweat Chloride at Week 24
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Data was reported as per the dose received and for overall participants.
Time Frame: Part B: Baseline, Week 24
Population: Part B Safety set included all participants who received at least 1 dose of study drug in part B. Number of participants analyzed is for participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Number analyzed (Participants) | 7 | 18 | 25
millimole per liter (mmol/L) | -47.07 (24.256) | -46.78 (27.584) | -46.86 (26.193)

5. Secondary Outcome: Part B: Absolute Change From Baseline in Weight at Week 24
Description: Data was reported as per the dose received and for overall participants.
Time Frame: Part B: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Number analyzed (Participants) | 9 | 24 | 33
kilograms (kg) | 1.00 (0.418) | 1.50 (0.552) | 1.36 (0.561)

6. Secondary Outcome: Part B: Absolute Change From Baseline in Stature at Week 24
Description: Stature was measured as height if children could stand unassisted and follow directions; otherwise, stature was measured as length. Data was reported as per the dose received and for overall participants.
Time Frame: Part B: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Number analyzed (Participants) | 9 | 23 | 32
centimeters (cm) | 2.5 (1.45) | 3.5 (0.93) | 3.3 (1.17)

7. Primary Outcome: Part A: Plasma Concentration of Ivacaftor and Its Metabolites
Description: Plasma concentration was reported for ivacaftor and its metabolites (hydroxymethyl ivacaftor [M1] and ivacaftor carboxylate [M6]) up to 24 hours post-dose on Day 4 (Hour 0 [pre-dose] on Day 1 and Day 4; 2, 3, 6, 24 hours post-dose on Day 4). Data was planned to be reported for overall participants in the period.
Time Frame: Part A: up to 24 hours post-dose on Day 4
Population: Part A Safety set included all participants who received at least 1 dose of study drug in part A.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: Overall Ivacaftor
Number analyzed (Participants) | 9
nanogram per milliliter (ng/mL)
  Ivacaftor: Hour 0 on Day 1 | 0.00 (0.00)
  Ivacaftor: Hour 0 on Day 4 | 396 (337)
  Ivacaftor: 2 Hours Post-Dose on Day 4 | 726 (284)
  Ivacaftor: 3 Hours Post-Dose on Day 4 | 957 (283)
  Ivacaftor: 6 Hours Post-Dose on Day 4 | 542 (241)
  Ivacaftor: 24 Hours Post-Dose on Day 4 | 124 (149)
  M1: Hour 0 on Day 1 | 0.00 (0.00)
  M1: Hour 0 on Day 4 | 1240 (723)
  M1: 2 Hours Post-Dose on Day 4 | 1540 (578)
  M1: 3 Hours Post-Dose on Day 4 | 2310 (820)
  M1: 6 Hours Post-Dose on Day 4 | 1580 (622)
  M1: 24 Hours Post-Dose on Day 4 | 389 (336)
  M6: Hour 0 on Day 1 | 0.00 (0.00)
  M6: Hour 0 on Day 4 | 1150 (709)
  M6: 2 Hours Post-Dose on Day 4 | 1050 (606)
  M6: 3 Hours Post-Dose on Day 4 | 1300 (614)
  M6: 6 Hours Post-Dose on Day 4 | 1390 (532)
  M6: 24 Hours Post-Dose on Day 4 | 439 (355)

8. Secondary Outcome: Part B: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI = (Weight [in kg]) divided by (Stature [in meters])^2. Data was reported as per the dose received and for overall participants.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Number analyzed (Participants) | 9 | 23 | 32
kilogram per square meter (kg/m^2) | 0.332 (0.5393) | 0.314 (0.5492) | 0.319 (0.5378)

ADVERSE EVENTS:
Time Frame: Part A: up to 93 days; Part B: up to 28 weeks
Description: Adverse events were reported separately for each part and as per the dose received and for overall participants in each part.
Arm/Group | Part A: Ivacaftor 50 mg | Part A: Ivacaftor 75 mg | Part A: Overall Ivacaftor | Part B: Ivacaftor 50 mg | Part B: Ivacaftor 75 mg | Part B: Overall Ivacaftor
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/9 | 3/10 | 3/24 | 6/34
Other Adverse Events (participants affected / at risk) | 3/4 | 5/5 | 8/9 | 9/10 | 23/24 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Ivacaftor 50 mg (N=4) | Part A: Ivacaftor 75 mg (N=5) | Part A: Overall Ivacaftor (N=9) | Part B: Ivacaftor 50 mg (N=10) | Part B: Ivacaftor 75 mg (N=24) | Part B: Overall Ivacaftor (N=34)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pseudomonas test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Ivacaftor 50 mg (N=4) | Part A: Ivacaftor 75 mg (N=5) | Part A: Overall Ivacaftor (N=9) | Part B: Ivacaftor 50 mg (N=10) | Part B: Ivacaftor 75 mg (N=24) | Part B: Overall Ivacaftor (N=34)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4 | 15 | 19
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 5 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2 | 5 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 3
Dysponea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nasal inflamation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory track congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 7 | 8
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 3
Gastroentritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Viral rash (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 3 | 6 | 9
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 3 | 3
Haemophilus test positive (Investigations) | 0 | 0 | 0 | 0 | 3 | 3
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1
Antibiotic resistant Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatic enzyme increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 4 | 4 | 2 | 6
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 1 | 1
Product taste abnormal (General disorders) | 0 | 1 | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 2
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Amblyopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anisometropia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.